CLINICAL TRIAL: NCT04908098
Title: Clinical and Biochemical Evaluation of the Effectiveness of Diode Laser Application With Non-Surgical Periodontal Treatment
Brief Title: Diode Laser Application With Non-Surgical Periodontal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ali Tugrul Gur, principal investigator, research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSA-2019-18111
Record Dates: First submitted 2021-05-08; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Periodontitis
Keywords: periodontitis; Gingival crevicular fluid; diode laser; sclerostin; TWEAK
MeSH Terms: conditions — Periodontitis; Sclerosteosis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups as study and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): Root-planning was performed using Gracey curettes in the areas where periodontal pockets were diagnosed after scaling. Laser application was then applied to the areas where root planning was applied. Laser was applied in continuous phase at 0.80W power, 940 nm wavelength and 0.80 J / s energy level.
  Interventions: Device: diode laser; Procedure: scaling - root planning
- Control group (Active Comparator): Root-planning was performed using Gracey curettes in the areas where periodontal pockets were diagnosed after scaling.
  Interventions: Procedure: scaling - root planning

INTERVENTIONS:
Device: diode laser — It is the application of the laser tip parallel to the inner surface of the periodontal pocket
  Arms: Laser group
Procedure: scaling - root planning — Scaling is the removal of calculus and other deposits in the root of the tooth.Root planning is the removal of necrotic cementum on the tooth root surface. Scaler and gracey curettes are used for these operations.

SUMMARY:
Periodontitis is an infectious disease that causes destruction of periodontal tissues with complex etiology that develops due to local and systemic factors. Host-derived enzymes, cytokines and proinflammatory markers are the main elements that play a role in this degradation. New techniques such as non-surgical or surgical methods combined with laser application are used for its treatment.

The subjects were divided into two groups as "Individuals Applied with Diode Laser in Addition to Non-Surgical Periodontal Treatment" (Laser group) and "Individuals with Non-Surgical Periodontal Treatment (SRP)" (Control group). While only non-surgical periodontal treatment was applied to individuals in the control group; In the laser group, diode laser was applied in addition to this treatment. All individuals were examined 1 and 3 months after treatment.The scaling root planing (SRP) procedure was performed mechanically with gracey curettes under local anesthesia. The diode laser applied to the study group was applied parallel to the gingival sulcus at 0.80W power, 940 nm wavelength and 0.80 J / s energy level in continuous phase. Gingival crevicular fluid (GCF) samples were taken without any procedure in order not to change the amount and content. All clinical parameters were also measured by the same investigator before SRP and in all participants. After this treatment, the participants were re-examined in the 1st and 3rd months for control purposes and GCF samples were taken from the same regions again and the clinical parameters were measured again by the same researcher. GCF samples were stored at -20 degrees Celsius until ELISA studies were performed. Clinical parameters (pocket depth, clinical attachment loss, bleeding on probing, gingival index, plaque index) and gingival crevicular fluid (GCF) sampling were obtained at each control. IL-1β, IL-10, IL-17, OPG, RANKL, TWEAK, Sclerostin levels in GCF samples were measured with ELISA method.

The aim of this study is to evaluate the effectiveness of diode laser application in addition to non-surgical treatment in periodontitis treatment clinically and biochemically and to assess the potential biomarkers for use.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of 5mm or more periodontal pockets on one or more surfaces in periodontal tissues,
2. Not having periodontal treatment in the last 3 months,
3. The informed consent form must be approved,
4. At least 18 years old.

Exclusion Criteria:

1. Presence of systemic disease,
2. Smoking,
3. Regular use of non-steroidal anti inflammatory drugs,
4. Having been treated with antibiotics in the last 3 months,
5. Individuals in need of pre-treatment antibiotic prophylaxis,
6. Pregnancy and lactation,
7. Not approving the informed consent form,
8. Patients with known allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study was the control examination performed 3 months after the first examination. At the 3rd month control, the same researcher measured clinical parameters from all patients | 3 months
  Probing depth is the measurement from the free gingival margin, to the base of the pocket in millimeters of the distance. Periodontal probe is used.

SECONDARY OUTCOMES:
The secondary outcome of the study is the recording of bleeding index in the 3rd month. | 3 months
  The bleeding index is evaluated as positive if there is bleeding in the gingiva during probing.
Another outcome of the study is the collection of gingival crevicular fluid samples in the 3rd month. | 3 months
  Samples are obtained by means of paper strips placed gently in the gingival groove. These samples are stored at -20 ° C for later analysis by ELISA method.
The secondary outcome of the study is a measure of the clinical attachment level. | 3 months
  The distance in millimeters from the cemento enamel junction to the bottom of the pocket.
The secondary outcome of the study is the recording of gingival index in the 3rd month. | 3 months
  The gingival index is graded as follows:
  0 = Normal gingiva
  1. = Mild inflammationslight change in color, slight oedema. No bleeding on probing
  2. = Moderate inflammation redness, oedema and glazing. Bleeding on probing
  3. = Severe inflammation marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.
The secondary outcome of the study is the recording of plaque index in the 3rd month. | 3 months
  The plaque index is graded as follows:
  0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Tuğrul Gür, Dentist, Principal Investigator — Principal Investigator; Güliz Nigar Güncü, Professor, Study Director — study director; Abdullah Cevdet Akman, professor, Principal Investigator — Study principal investigator; Rahime Meral Nohutcu, professor, Principal Investigator — study principal investigator; Aslı Pınar, Professor, Principal Investigator — biochemistry
Locations (1):
- Hacettepe Universty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual data of the participants will not be shared. Statistical analysis of the study will be shared.